CLINICAL TRIAL: NCT05289440
Title: The Effect of Esketamine on the Quality of Recovery After Modified Radical Mastectomy
Brief Title: Esketamine Administration on Recovery Quality After Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Zhumin
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Esketamine and the Quality of Recovery
Keywords: Esketamine; The quality of recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose esketamine infusion on the quality of recovery after radical mastectomy (Experimental): Patients received a bolus infusion of esketamine (0.5 mg/kg) before cutting the skin, and then esketamine was infused at a rate of 2 µg/kg/min until before suture the skin.
  Interventions: Drug: Low-dose esketamine infusion; Drug: High-dose esketamine infusion; Drug: Saline infusion
- High-dose esketamine infusion on the quality of recovery after radical mastectomy (Experimental): Patients received a bolus infusion of esketamine (0.5 mg/kg) before cutting the skin, and then esketamine was infused at a rate of 4 µg/kg/min until before suture the skin.
  Interventions: Drug: Low-dose esketamine infusion; Drug: High-dose esketamine infusion; Drug: Saline infusion
- Saline infusion on the quality of recovery after radical mastectomy (Experimental): Patients received a bolus infusion of the same volume saline before cutting the skin, and then the same volume saline was infused until before suture the skin.
  Interventions: Drug: Low-dose esketamine infusion; Drug: High-dose esketamine infusion; Drug: Saline infusion

INTERVENTIONS:
Drug: Low-dose esketamine infusion — Patients received a bolus infusion of esketamine (0.5 mg/kg) before cutting the skin, and then esketamine was infused at a rate of 2 µg/kg/min until before suture the skin.
Drug: High-dose esketamine infusion — Patients received a bolus infusion of esketamine (0.5 mg/kg) before cutting the skin, and then esketamine was infused at a rate of 4 µg/kg/min until before suture the skin.
Drug: Saline infusion — Patients received a bolus infusion of the same volume saline before cutting the skin, and then the same volume saline was infused until before suture the skin.

SUMMARY:
Some studies have reported that intravenous esketamine reduce postoperative pain intensity. The investigators investigated whether esketamine could improve the the quality of recovery after modified radical mastectomy.

DETAILED DESCRIPTION:
A total of 111 patients were randomly allocated into 3 groups. Patients in group LE received a bolus infusion of esketamine (0.5 mg/kg) before cutting the skin, and then esketamine was infused at a rate of 2 µg/kg/min until before suture the skin. Patients in group HE received a bolus infusion of esketamine (0.5 mg/kg) before cutting the skin, and then esketamine was infused at a rate of 4 µg/kg/min until before suture the skin. Patients in group CON received a bolus infusion of the same volume saline before cutting the skin, and then the same volume saline was infused until before suture the skin.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status
* Scheduled for elective modified radical mastectomy

Exclusion Criteria:

* Severe respiratory disease
* Renal or hepatic insufficiency
* History of preoperative psychiatric
* Preoperative hypertension
* Preoperative history of chronic pain

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Quality of recovery scores (QoR-15) | 1 day after operation
  Our primary outcome was quality of recovery scores (QoR-15) 1 day after operation

SECONDARY OUTCOMES:
Pain visual analogue scale scores | The first 48 hours after operation
  Secondary Outcome Measure was pain visual analogue scale scores

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anqing Hospital Anesthesiology, Anqing, Anhui, China